CLINICAL TRIAL: NCT03935945
Title: Personalized Feedback to Reduce HIV+ Hazardous Drinking in Primary Care
Brief Title: Brief Personalized Feedback Intervention for Hazardous Drinking in an HIV Clinic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Clayton Neighbors, Moores Professor and Director of Social Psychology Program, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: uhouston
Record Dates: First submitted 2018-01-10; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-05

CONDITIONS: Alcohol Consumption
Keywords: Drinking; Alcohol; HIV+
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Feedback Intervention (PFI) (Experimental): Participants in the intervention group will receive a computerized personalized feedback intervention (PFI) lasting approximately 20-30 minutes.
  Interventions: Behavioral: Personalized Feedback Intervention
- Attention-Control (No Intervention): Attention control information will be comparable in focus on health-related behaviors (e.g., nutrition, exercise). We will use behaviors in the attention control feedback that are not associated with study outcomes. Attention control feedback will have text and graphs that are similar in appearance and length (i.e., 20-30 minutes) to intervention feedback.

INTERVENTIONS:
Behavioral: Personalized Feedback Intervention — Participants in the intervention group will receive a computerized personalized feedback intervention (PFI) lasting approximately 20-30 minutes. PFI highlights discrepancies between one's own drinking and typical drinking; reframes use in terms of personal, social, financial, and health consequences; and, offers strategies for reducing alcohol use. The feedback is non-confrontational in tone, seeks to increase motivation to reduce drinking and is based on the information provided during the baseline assessment
  Arms: Personalized Feedback Intervention (PFI)

SUMMARY:
The objective of the proposed research is test the feasibility of a brief computer-based personalized feedback intervention to reduce heavy alcohol use among HIV+ individuals. There is a critical need to develop accessible, empirically-supported, low-threshold interventions for HIV+ hazardous alcohol users. The proposed research will develop and evaluate the feasibility, acceptability, and potential efficacy of a novel evidence- and computer-based Personalized Feedback Intervention (PFI) among HIV+ hazardous alcohol users in a high volume Houston HIV clinic.

H1: The PFI group will show increases in self-efficacy, intention to reduce or quit drinking, and decreases in actual drinking, relative to the control group.

H2: Reduced drinking will be associated with less risky sexual behavior, better antiretroviral therapy (ART) medication adherence, and improved HIV quality of life.

H3: Changes in normative perceptions, alcohol use attitudes, self-efficacy for alcohol abstinence, intentions to use, alcohol outcome expectancies, and protective behavioral strategies will mediate intervention effects on drinking behavior. Even if the investigators do not find significant effects on our main outcomes, these will also serve as useful proximal dependent variables that will provide important information regarding the feasibility of this intervention approach in this population.

H4: Intervention effects on drinking outcomes will be stronger for those who report drinking more for social and/or coping reasons.

DETAILED DESCRIPTION:
The objective of the proposed research is test the feasibility of a brief computer-based personalized feedback intervention to reduce heavy alcohol use among HIV+ individuals. Rates of hazardous alcohol use among HIV+ individuals are approximately two times that found in the general population. Hazardous alcohol use contributes to problems with HIV medication adherence, risky sexual behavior, and psychological problems, as well as physical complications (rapid disease progression, medication toxicities, organ failure, and poor viremic control), which may lead to increased risk of transmission and premature death. Yet, HIV+ hazardous alcohol users remain a hard-to-reach and underserved group. There is therefore a critical need to test alternative approaches to the implementation of effective interventions to reduce HIV disease transmission and progression in HIV+ hazardous alcohol users. One novel and promising intervention approach is the use of personalized feedback, which has consistently been found to be efficacious for reducing hazardous alcohol use across a number of populations. Personalized feedback highlights discrepancies between one's own drinking and typical drinking; reframes use in terms of personal, social, financial, health, and other consequences; and offers strategies for reducing use and alcohol-related negative consequences. The proposed research will develop and evaluate the feasibility, acceptability, and potential efficacy of a novel evidence- and computer-based Personalized Feedback Intervention (PFI) among HIV+ hazardous alcohol users in a high volume Houston HIV clinic. The investigators will recruit 150 HIV+ hazardous alcohol users randomly assigned to receive either PFI or attention-control feedback (e.g., diet, exercise). The investigators expect to demonstrate feasibility and acceptability of the PFI. Outcomes include drinking change processes and behavior, alcohol-related risky sexual behavior, and HIV-related outcomes. An underlying premise, which will be evaluated through the aims, is that the difficulty in reaching hazardous alcohol users who are HIV+ can be addressed with an approach that will not be burdensome to the individuals or to clinic staff. All assessments and procedures will take place in the clinic on tablets or laptop computers. Follow-up assessments will occur at 3 months post-baseline. This research builds on the collaborative work of an experienced team of investigators with complementary expertise supporting all aspects of the proposed research.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ as confirmed by medical records
* AUDIT scores for the last 30 days to be ≤7 for women and ≤8 for men
* Between the ages of 18 and 50
* Not currently pregnant
* Reading level on Word Reading component of Wide Range Achievement Test (WRAT-4) at or above a 5th grade level and proficient in English (although English does not have to be the first language, they must be fluent enough to understand study materials and measures)
* Not currently in alcohol treatment
* Do not have a current psychiatric diagnosis that would preclude them from being in our study as determined by the MINI (MINI INTERNATIONAL NEUROPSYCHIATRIC INTERVIEW) neuropsychiatric interview

Exclusion Criteria:

* Not meeting inclusion criteria
* Unwillingness to participate
* Failure to provide consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-01-20 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
Typical weekly drinking | Change from baseline to 3-month follow-up
  Typical weekly drinking will be measured with the Daily Drinking Questionnaire (DDQ), which asks how much a person drinks on a typical day of each week, for the past 3 months. Drinks will be measured by standard drinks. The scale ranges from 0 drinks to 25 drinks per day (leading to a maximum for 175 weekly drinks).
Quantity of Alcohol Consumed in Single Occasion | Change from baseline to 3-month follow-up
  This involves the number of drinks consumed in a single occasion in the past month. This outcome will be measured by the change in responses of Quantity-Frequency-Peak Alcohol Use Index (QF) between baseline and 3-month follow-up.
Problematic Drinking | Change from baseline to 3-month follow-up
  This outcome looks at the amount of alcohol consumed and any alcohol-related consequences as a result of participant drinking. This outcome will be measured by the change in responses of the Alcohol Use Disorders Identification Test (AUDIT) between baseline and 3-month follow-up.
Consequences | Change from baseline to 3-month follow-up
  This outcome looks at any consequences related to drinking. This outcome will be measured by the change in responses of the Drinker Inventory of Consequences (DRINC) between baseline and 3-month follow-up.

SECONDARY OUTCOMES:
Sexual behavior | Change from baseline to 3-month follow-up
  Sexual behavior will be assessed with questions about sex partners, unprotected sex, vaginal/anal sex, sex with alcohol will be assessed via the Sexual Behavior and Alcohol-Related Sexual Behavior questionnaire, a questionnaire previously used by Dr. Lewis that is well-validated and has been used in her prior NIH funded work. The Alcohol-Related Sexual Behavior questionnaire ranges from none to 25+ times for the amount of time that participants engaged in sex in the past 3 months.
Alcohol-related sexual behavior | Change from baseline to 3-month follow-up
  Sex with alcohol will be assessed via the Sexual Behavior and Alcohol-Related Sexual Behavior questionnaire, a questionnaire previously used by Dr. Lewis that is well-validated and has been used in her prior NIH funded work. The Alcohol-Related Sexual Behavior questionnaire ranges from none to 25+ times for alcohol use in conjunction with oral, vaginal, or anal sex.
Medication Adherence | Change from baseline to 3-month follow-up
  Medication adherence will be measured using self-report (ACTG questionnaire), which asks questions as to a patient's medication adherence from a scale of 0 (not at all) to 3 (extremely sure).
Viral load measures | Change from baseline to 3-month follow-up
  Viral load measures will be determined through chart review with permission from the research participant.
Unannounced pill counts | Change from baseline to 3-month follow-up
  Unannounced pill counts will provide an objective measure of adherence that is significantly associated with other measures of adherence including electronic monitors.
Quality of Life | Change from baseline to 3-month follow-up
  We will also assess HIV-related quality of life with the validated World Health Organization (WHO) HIV Quality of Life measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong CCY, Paulus DJ, Lemaire C, Leonard A, Sharp C, Neighbors C, Brandt CP, Lu Q, Zvolensky MJ. Examining HIV-Related stigma in relation to pain interference and psychological inflexibility among persons living with HIV/AIDS: The role of anxiety sensitivity. J HIV AIDS Soc Serv. 2018;17(1):1-15. doi: 10.1080/15381501.2017.1370680. Epub 2017 Nov 30. PMID 30034300
- [Background] Paulus DJ, Jardin C, Bakhshaie J, Sharp C, Woods SP, Lemaire C, Leonard A, Neighbors C, Brandt CP, Zvolensky MJ. Anxiety sensitivity and hazardous drinking among persons living with HIV/AIDS: An examination of the role of emotion dysregulation. Addict Behav. 2016 Dec;63:141-8. doi: 10.1016/j.addbeh.2016.07.013. Epub 2016 Jul 21. PMID 27497249
- [Background] Wong CCY, Paulus DJ, Lemaire C, Leonard A, Sharp C, Neighbors C, Brandt CP, Zvolensky MJ. Emotion Dysregulation: An Explanatory Construct in the Relation Between HIV-Related Stigma and Hazardous Drinking among Persons Living with HIV/AIDS. Stigma Health. 2019 Aug;4(3):293-299. doi: 10.1037/sah0000113. Epub 2018 Jun 7. PMID 31777759
- [Background] Brandt CP, Jardin C, Sharp C, Lemaire C, Zvolensky MJ. Main and interactive effects of emotion dysregulation and HIV symptom severity on quality of life among persons living with HIV/AIDS. AIDS Care. 2017 Apr;29(4):498-506. doi: 10.1080/09540121.2016.1220484. Epub 2016 Aug 20. PMID 27546879

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT03935945/Prot_SAP_000.pdf